CLINICAL TRIAL: NCT00540332
Title: A Phase 1/2 Study to Evaluate Safety, Pharmacokinetics and Preliminary Efficacy of Weekly Doses of Palifermin (Recombinant Human Keratinocyte Growth Factor, rHuKGF) for the Reduction of Oral Mucositis in Subjects With Locally Advanced Head and Neck Cancer (HNC) Receiving Postoperative Radiotherapy
Brief Title: A Study of Palifermin for the Reduction of Oral Mucositis in Subjects With Locally Advanced Head and Neck Cancer Receiving Postoperative Radiotherapy
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The 20070201 study was terminated based on evaluation of Palifermin solid tumor data.
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Clinical Development, Biovitrum AB (publ)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 20070201; NCT00965159 (obsolete NCT alias)
Record Dates: First submitted 2007-10-04; First posted 2007-10-08 (Estimated); Last update posted 2009-03-02 (Estimated); Status verified 2009-01

CONDITIONS: Head and Neck Cancer
Keywords: Oncology; KGF; HNC; head and neck; oral mucositis; OM; proteinurea; palifermin; clinical trial
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms; Stomatitis | interventions — Fibroblast Growth Factor 7

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): Approximately 17 subjects to receive palifermin. Subjects will be enrolled as follows:
  * PK cohort will be randomized in a 3:1 ratio [palifermin: placebo] in at least 12 subjects
  * Non-PK cohort will be randomized in a 1:1 ratio [palifermin: placebo] in up to 28 subjects.
  Interventions: Drug: Placebo
- Palifermin (Experimental): Approximately 23 subjects to receive palifermin. Subjects will be enrolled as follows:
  * PK cohort will be randomized in a 3:1 ratio [palifermin: placebo] in at least 12 subjects
  * Non-PK cohort will be randomized in a 1:1 ratio [palifermin: placebo] in up to 28 subjects.
  Interventions: Drug: palifermin

INTERVENTIONS:
Drug: Placebo — Single IV dose of placebo, 3 days before the start of RT, then once weekly placebo doses at the same dose during a planned 6 week RT course.
  Arms: Placebo
Drug: palifermin — 120μg/kg, single IV, 3 days before the start of Radiotherapy (RT), then once weekly at the same dose during a planned 6-week RT course
  Arms: Palifermin

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of palifermin on the incidence of oral mucositis in subjects with locally advanced head and neck cancer receiving postoperative radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* History of newly diagnosed histologically confirmed squamous cell carcinoma (AJCC Stage II, III or IVA) involving either the oral cavity, oropharynx, hypopharynx, larynx and post surgical resection (R0 or R1)
* Candidates for postoperative RT-only treatment and scheduled to receive RT within 12 weeks of surgery
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Urinary protein-creatinine ratio (random sample, spot PCR) ≤ 0.2 mg/mg

Exclusion Criteria:

* Tumors of the lips, paranasal sinuses, salivary glands, or of unknown primary tumors and R2 resection margins
* Metastatic disease (M1)
* Presence or history of any other primary malignancy, other than curatively treated in situ cervical cancer, or basal cell carcinoma of the skin without evidence of disease for > 3 years
* History of pancreatitis
* Prior radiotherapy to the site of disease
* Prior chemotherapy or requiring chemotherapy during treatment phase of study
* Prior treatment with palifermin, or other fibroblast or keratinocyte growth factors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent proteinuria | 11 weeks
Duration of treatment-emergent proteinuria | 11 weeks
Incidence of chronic proteinuria | 11 weeks
Time (days) to onset of treatment-emergent proteinuria | 11 weeks
Maximum protein-to-creatinine ratio values during the treatment period | 11 weeks
Pharmacokinetic profile to include Systemic clearance, volume of distribution at steady state, estimated initial concentration, area under the conc-time curve, terminal half-life and mean residual time | in Week 1

SECONDARY OUTCOMES:
Time (days) to onset of severe Oral Mucositis WHO grade 3 or 4 | 11 weeks
Disease status at End of Treatment visit | 11 weeks
Incidence of serum anti-palifermin antibody formation | 11 weeks
Incidence of second primary tumors | up to 10 years (Long-Term Follow-Up phase)
Incidence of other malignancies | up to 10 years (Long-Term Follow-Up phase)
Progression-free survival | up to 10 years (Long-Term Follow-Up phase)
Overall survival | up to 10 years (Long-Term Follow-Up phase)
Incidence of adverse events and laboratory abnormalities | 11 weeks
Incidence (%) and duration (days) of severe Oral Mucositis WHO grade 3 or 4 | 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Biovitrum AB (publ)

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com